CLINICAL TRIAL: NCT04112147
Title: A Randomized, Double-Blind, Dosing-Ranging, Placebo-controlled Trial of Antroquinonol in Patients With Chronic Hepatitis B
Brief Title: A Randomized, Placebo-controlled Trial of Antroquinonol in Patients With Chronic Hepatitis B
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cheng-Chung Wei (Other)
Collaborators: Golden Biotechnology Corporation (Industry)
Responsible Party: Sponsor-Investigator, Cheng-Chung Wei, Chung Shan Medical University Hospital, Chung Shan Medical University
Organization: Chung Shan Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CS18018
Record Dates: First submitted 2019-10-01; First posted 2019-10-02 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-10

CONDITIONS: Chronic Hepatitis B
Keywords: antroquinonol, Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — antroquinonol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Antroquinonol capsule 100mg (Experimental): Patients will receive 12-week of 50mg BID Antroquinonol
  Interventions: Drug: Antroquinonol capsule 100mg
- Antroquinonol capsule 200mg (Experimental): Patients will receive 12-week of 100mg BID Antroquinonol
  Interventions: Drug: Antroquinonol capsule 200mg
- Placebo oral capsule (Placebo Comparator): Patients will receive 12-week of 50mg BID Antroquinonol placebo
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Antroquinonol capsule 100mg — Patients will receive 12-week of 50mg BID Antroquinonol
  Other Names: Antroquinonol 100mg
  Arms: Antroquinonol capsule 100mg
Drug: Antroquinonol capsule 200mg — Patients will receive 12-week of 100mg BID Antroquinonol
  Other Names: Antroquinonol 200mg
  Arms: Antroquinonol capsule 200mg
Drug: Placebo oral capsule — Patients will receive 12-week of 100mg BID Antroquinonol placebo
  Other Names: Placebo
  Arms: Placebo oral capsule

SUMMARY:
Primary Objective:

To evaluate the activity of Antroquinonol in patients with chronic hepatitis B

Secondary Objective:

To assess the mechanism and cytokines change of Antroquinonol in patients with chronic hepatitis B

DETAILED DESCRIPTION:
This is a Phase II, three-arms, double-blind, dosing-ranging, placebo-controlled trial evaluating the efficacy of Antroquinonol in patients with chronic hepatitis B. The study is conducted in compliance with the guidelines for Good Clinical Practice and the Declaration of Helsinki. Approval is obtained from the local ethics committee or institutional review board at each study center. All the patients provided written informed consent.

60 patients totally (20 patients per arm) with chronic hepatitis B will receive Antroquinonol or placebo. A patient will have received at one dose of Antroquinonol or placebo. Enrollment will continue until the target number of evaluable patients has been enrolled.

Written informed consent must be obtained from all patients before initiating Screening. The Screening period will be up to 14 days in duration (Days -14 to -1). Following completion of all Screening assessments and confirmation of eligibility criteria, patients will receive Antroquinonol 100mg, 200mg or placebo per day on Day 1 for 12 weeks or until documented evidence of virus DNA > 10 x [minimum], unacceptable toxicity, non-compliance or withdrawal of consent by the patient, or the investigator decides to discontinue treatment, whichever comes first. The time of study drug administration should be recorded in the patient diary.

Patients will attend study visits on Days 1, 29, 57 and 85. The following procedures will be performed according to the schedule of assessments: physical examination, vital signs, clinical laboratory tests, adverse events (AEs), concomitant medication and patient compliance.

The primary endpoint is the change from baseline in quantitative hepatitis B surface antigen (Log qHBsAg) at Day 85.

ELIGIBILITY:
Inclusion criteria -

1. Chronic HBV infection patients between the ages of 20 and 75 years with serum hepatitis B surface antigen(HBsAg) positivity for more than 6 months
2. BMI≦35
3. HBsAg≧10 IU/mL and HBV DNA≧2000 IU/mL.
4. GOT or GPT ≧ 25 IU
5. Female subject must use effective methods of contraception
6. No abnormal finding of clinical relevance
7. Written informed consent

Exclusion criteria -

1. Evidence of hepatic decompensation such as:

   1. Coagulopathy defined as prolongation of prothrombin time greater than 3 seconds
   2. Total bilirubin of 2 times the upper limit of normal
   3. FIB-4 of 3.25 or greater
2. Abnormal hematological and biochemical parameters at screening

   1. White blood cell count less than 2500 cells/uL
   2. Absolute neutrophil count (ANC) less than 1,000 cells/mm3 (less than 750 mm3 for African or African-American subjects)
   3. Hemoglobin less than 12 g/dL for males, less than 11 g/dL for females
   4. Estimated GFR less than 50 mL/min
3. Suspected or confirmed liver diseases from etiologies other than HBV (such as alcohol, toxin, drug, shock, acute viral hepatitis A or E), co-infection with human immunodeficiency virus, hepatitis C virus or hepatitis delta virus, prior antiviral treatment with NUCs or interferon, and recent immunosuppressive therapy (including chemotherapy and systemic corticosteroid).
4. Immunodeficiency disorders or severe autoimmune disease
5. Severe pulmonary disorders or significant cardiac diseases
6. Gastrointestinal disorder with post-operative condition that could interfere with drug absorption
7. Significant psychiatric illness that in the judgment of the Investigator, is a contraindication to protocol participation or impairs a volunteer's ability to give informed consent
8. Any malignancy diagnosed within 5 years or evidence of hepatocellular carcinoma (e.g., α fetoprotein > 50ng/mL or radiologic evidence)
9. Solid organ transplantation
10. Current drug or alcohol abuse
11. Pregnancy or lactation
12. Under hepatitis B antiviral or interferon treatment within 3 months

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-08-10 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
quantitative hepatitis B surface antigen (Log qHBsAg) | Week 0 and Week 12
  The primary endpoint is the change from baseline in quantitative hepatitis B surface antigen (Log qHBsAg) at Week 12.

SECONDARY OUTCOMES:
serum hapatitis B virus DNA level | Week 0, Week 4, Week 8 and Week 12
  Change from baseline serum hapatitis B virus DNA level(HBV DNA as measured in IU/mL) at Week 4, Week 8 and Week 12
hepatitis B surface antigen | Week 0, Week 4 and Week 8
  Change from baseline quantitative hepatitis B surface antigen at Week 4 and Week 8
Fibrosis-4(FIB-4) scale | Week 0 and Week 12
  Changes from baseline FIB-4 scale at Week 12
Hepatitis B surface antigen loss (HBeAg loss) | Week 12
  Percentage of HBeAg loss at Week 12
glutamate oxaloacetate transaminase (GOT) | Week 0 and Week 12
  Change from baseline GOT at Week 12
Glutamic Pyruvic Transaminase (GPT) | Week 0 and Week 12
  Change from baseline GPT at Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Wei C- C, M.D., Principal Investigator — Chung Shan Medical University
Locations (1):
- Chung Shan Medical University hospital, Taichung, Taiwan